CLINICAL TRIAL: NCT04577378
Title: Efficacy and Safety of Drug Combination Therapy of Isotretinoin and Some Antifungal Drugs as A Potential Aerosol Therapy for COVID-19 : An Innovative Therapeutic Approach
Brief Title: Efficacy and Safety of Drug Combination Therapy of Isotretinoin and Some Antifungal Drugs as A Potential Aerosol Therapy for COVID-19 : An Innovative Therapeutic Approach COVID-19
Acronym: Isotretinoin
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Mahmoud Ramadan mohamed Elkazzaz, Principal Investigator, Kafrelsheikh University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: Isotretinoin
Record Dates: First submitted 2020-04-13; First posted 2020-10-06 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Patients and method :
  13- This study will performed on 45 patients tested positive for the presence of COVID-19 RNA by RT-PCR kit for RNA detection will randomly divided into 3 equal groups
Who Masked: Participant
Masking Description: Single (Participant)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- 13 cis retinoic acid doses orally (Active Comparator): The infected patients will receive Aerosolized 13 cis retinoic acid in gradual in one dose per day increases from 0.2 mg/kg/day to 4 mg/kg/day as inhaled 13 cis retinoic acid therapy for 14 days plus aerosolized Itraconzaole powder: single dose of 5mg/kg/day for 14 days
  Interventions: Drug: Drug: Isotretinoin(Aerosolized 13 cis retinoic acid) plus Aerosolized Itraconazole
- Aerosolized 13 cis retinoic acid (Sham Comparator): The infected patients will receive Aerosolized 13 cis retinoic acid in gradual in one dose per day increases from 0.2 mg/kg/day to 4 mg/kg/day as inhaled 13 cis retinoic acid therapy for 14 days plus Aerosolized Itraconzaole powder: single dose of 5mg/kg/day for 14 days
  Interventions: Drug: Drug: Isotretinoin(Aerosolized 13 cis retinoic acid)
- control (No Intervention): No intervention

INTERVENTIONS:
Drug: Drug: Isotretinoin(Aerosolized 13 cis retinoic acid) plus Aerosolized Itraconazole — After randomization, erosolized 13 cis retinoic acid in gradual one dose increases froms 0.2 mg/kg/day to 4 mg/kg/day as inhaled 13 cis retinoic acid therapy for 14 days plus Aerosolized Itraconazole 5mg per day for 14 days
  Arms: 13 cis retinoic acid doses orally
Drug: Drug: Isotretinoin(Aerosolized 13 cis retinoic acid) — Drug: Aerosolized 13 cis retinoic acid in gradual one dose increases froms 0.2 mg/kg/day to 4 mg/kg/day as inhaled 13 cis retinoic acid therapy for 14 days
  Arms: Aerosolized 13 cis retinoic acid

SUMMARY:
Efficacy and safety of Drug combination therapy of Isotretinoin and some Anti fungal Drugs as A potential Aerosol therapy for COVID-19 : An innovative therapeutic approach

The pandemic of COVID-19 which is caused by severe acute respiratory syndrome coronavirus 2 (SARS-COV-2) has infected over 2,000,000 people causing over 150,000 deaths.It hasno currently approved treatments.. Airborne SARS-CoV-2 infections in humans initiate from the virus entering nasal and airway epithelial cells through binding to angiotensin-converting enzyme 2 (ACE2). TMPRSS2, a cellular protease that activates the SARS-CoV-2 spike protein, colocalizes with ACE2 and can prime SARS-CoV-2 fusion directly at the plasma membrane. In the lungs, SARS-CoV-2 infects type I and type II alveolar epithelial cells, as well as alveolar macrophages that are among the first producers of pro-inflammatory cytokines. As key components of the immediate antiviral response, type I interferons (here after referred to as IFNs) are crucial for restricting viral replication and spread, through autocrine and paracrine type I IFN receptor (IFNAR) signalling. However, minimal amounts of IFNs have been detected in the peripheral blood or lungs of patients with severe COVID-19 In a mouse model of SARS-CoV infection, local IFN responses in the lungs were delayed relative to peak viral replication, which impeded virus clearance and was associated with the development of CRS . SARS-CoV-2 ORF3b is a potent interferon inhebitor and antagonist Here, we review the molecular mechanisms by which Retinoic acid (isotretinoin) and antifungal drugs can cooperate to induce interferon in covid-19 infected patients A study reported that 13 Cis retinoic acid induced significant upregulation of toll-like receptor 3 resulting in an immune response to dsRNA intermediate which can be partially generated during CoV-2 replication . TLR3 sensitized by dsRNA and cascades of signaling pathways (Interferon-regulatory factor 1 (IRFs) and Nuclear factor-κB (NFκB) activation, respectively) are activated to produce type I interferons. The production of type I IFNs is important to enhance the release of antiviral proteins for the protection of uninfected cells. RA can be generated in multiple forms as all-trans, 9-cis,and 13-cis retinoic acid. A study reported that Retinoic acid induces directly the expression of two transcription factors, Stat1 and IRF-1 which play central roles in the IFN signal transduction. In addition, RA induces IFN-a synthesis, IFNs can serve as the first line of immune defense against viral infections. IFNs are very powerful cytokines, which play a key role in combatting pathogenic infections by controlling inflammation and immune response by directly inducing antipathogen molecular countermeasures. There are three classes of IFNs: type I, type II, and type III. Antifungal drug. Fluconazol or itraconazol can inhibit cytochrome P450 enzymes, especially cype 26 which control retinoic acid concentration into human cells enhance both isotretinoin effect and Concentrations in Target Tissues This in turn lead to hyper interferon induction and synthesis in case of COVID-19. Also a study demonstrated that isotretinoin can be given as aerosolized via inhalation rout without any damage in lung cells. Repeated high doses of 13 cis retinoic by inhalation resulted in moderate loss of body weight, but microscopic investigation of ten tissues including lung and oesophagus did not detect any significant aerosol-induced damage therefore inhaled isotretinoin might provide sufficient drug to the target cells in lung for efficacy while avoiding systemic toxicity. In conclusion,isotretinoin therapy has furthermore a proven anti-inflammatory, anti-platelet and fibrinolytic activities which may protect patients infected with covid-19 from widespread blood clots. From this point, we suggest that isotretinoin will be the immunity passport" in the context of COVID-19.

DETAILED DESCRIPTION:
This is a small pilot study investigating whether there is any efficacy signal of combination therapy of Isotretinoin and some Anti fungal Drugs in COVID-19 treatment that warrants a larger Phase III trial, or any harm that suggests that such a trial should not be done. It is expected to produce statistically significant results in the major endpoints. The investigator will examine all of the biologic, physiological, and clinical data to determine whether a Phase III trial is warranted.

Primary efficacy analysis will be carried only on patients receiving at least 4 doses of active combination drug. Safety analysis will be carried out on all patients receiving at least one dose of active drug.

introduction

In Wuhan, Hubei Province, China, cases of acute respiratory infection were reported in December 2019.1,2 The Chinese Center for Disease Control and Prevention (CDC), initially reported that the cause of this disease is severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), then it is founded to be a novel coronavirus.3Now, This disease, is designated by the WHO as coronavirus disease 2019 (COVID-19), which rapidly spreads to other cities of China, and has become a public health emergency of international concern (PHEIC) following its global spread. The clinical manifestations of COVID-19 are fever, cough, muscle pain, fatigue, diarrhea and pneumonia, and can cause death in severe cases.4China has reported 72436 cases of confirmed COVID-19 and 1868 fatalities through February 18, 2020.5 The innate immune system represents the first line of defense and initiates counteractive responses that protect the host from viral infection through evolutionarily conserved pattern recognition receptors (PRR) 6. PRRs include the membrane-bound Toll-like receptors (TLRs) and cytosolic sensors, such as retinoic acidinducible gene-I (RIG-I)-like receptors (RLRs), which sense RNA viruses 6. RIG-I specifically detects the intracellular double-stranded viral RNA bearing 5' triphosphate and panhandle structures to activate antiviral signaling7,8. Once a host is invaded by a virus, PRRs transmit signals to the downstream kinases that activate transcription factors, including IFN regulatory factor-3 (IRF3), nuclear factor κB (NF-κB), and ATF-2/c-jun, with the help of different adaptor molecules (MAVS/IPS-1/VISA/Cardif for RIG-I, TRIF for TLR3, and MyD88 for TLR7/8/9) to activate IFN production9,10,11.Viruses have evolved elaborate mechanisms to evade or inactivate the innate immune signaling pathway for their replication 12. Severe acute respiratory syndrome (SARS) is a highly contagious respiratory disease that appeared first in China in 2002 and has infected more than 8000 people worldwide and killed about 800 of those infected. SARS coronavirus (SARS-CoV) has a singlestranded, positive sense RNA genome of approximately 29.7 kb 13,14. Numerous studies have revealed that SARS-CoV develops an antagonistic mechanism to evade the antiviral activities of IFN 15 Infection with SARS-CoV-2 can lead to excessive production of pro-inflammatory cytokines, but the production of type I interferons, which are key antiviral mediators, is reportedly blunted; Previous studies suggested that SARS-CoV papain-like protease (PLpro) inhibits activation of the IRF3 pathway, which would normally elicit a robust IFN response, but the mechanism(s) used by SARS PLpro to inhibit activation of the IRF3 pathway is not fully known.16 As key components of the immediate antiviral response, type I interferons are crucial for restricting viral replication and spread, through autocrine and paracrine type I IFN receptor (IFNAR) signalling. Type 1 interferons have a broad antiviral activity in vitro and are currently evaluated in a clinical trial to treat MERS-CoV However, minimal amounts of IFNs have been detected in the peripheral blood or lungs of patients with severe COVID-19 17,18 In a mouse model of SARS-CoV infection, local IFN responses in the lungs were delayed relative to peak viral replication, which impeded virus clearance and was associated with the development of CRS19 . SARS-CoV-2 ORF3b is a potent interferon inhebitor and antagonist 20 The dysregulated IFN responses are indicative of the effective immunomodulatory strategies used by betacoronaviruses. During the incubation phase, SARS-CoV-2 replicates stealthily in host cells without detectably triggering IFNs, leading to high viral loads1. Coronaviruses are known to induce the formation of membranous compartments dedicated to viral RNA synthesis and thereby conceal viral pathogen-associated molecular patterns (PAMPs; for example, viral RNAs) from detection by host pattern recognition receptors (PRRs), such as RIG-I and MDA5. Furthermore, several conserved betacoronavirus proteins, predominantly non-structural proteins (nsps), are known to exert direct IFN-antagonistic activities. Some modify specific features of the viral RNA (by catalysing guanosine-N7 and ribose-2'-O methylation) to avoid recognition by specific PRRs (for example, nsp14 and nsp16), while others, such as nsp3 and nsp1, inhibit the signal transduction mediated by PRRs and by IFNAR, respectively19

--Impact of TLR3 on type I IFNs

Toll-like receptors (TLRs) are a class of pattern recognition receptors (PRRs) that initiate innate immune response to invading pathogens by sensing conserved molecular patterns for early immune recognition of a pathogens like viruses, bacteria, and fungi to initiate innate immune response to invading pathogens . In addition ,TLRs play an important role in tissues repair and tissues injury- induced inflammation. The emergence of highly pathogenic severe acute respiratory syndrome coronaviruses (MERSCoV) is a concern for global public health, as there is a lack of efficacious vaccine platforms and antiviral therapeutic strategies21. A study demonstrated that pre-stimulation of TLR3 polyinosini- polycytidylic acid (poly I:C) hindered MHV infection through induction of INF- β in macrophages 22 A study demonstrated that TLR3(-/-), TLR4(-/-), and TRAM(-/-) mice are more susceptible to SARS-CoV than wild-type mice but experience only transient weight loss with no mortality in response to infection. In contrast, mice deficient in the TLR3/TLR4 adaptor TRIF are highly susceptible to SARS-CoV infection, showing increased weight loss, mortality, reduced lung function, increased lung pathology, and higher viral titers In further research, Tsai .and Chen showed the high level of IFN-α/β produced from the TLR3-IRF3/IRF7 pathway and IFN-β is the reason for inhibiting DENV replication. In HUH-7 cells, huTLR3 can recognize DENV-1 and induce the expression of IFN-β, which can enhance the expression of huTLR3 on the contrary . TLR3 also induces type I IFN during WNV..21

--Impact of isotretinoin 13 cis retinoic acid on TLR3 and TLR-2

Many of the significantly up-regulated genes are known to be retinoid-responsive genes including: retinoic acid responder 1 [tazarotene induced gene 1 (TIG1)}, cellular retinol binding protein 1 and cellular retinoic acid binding protein 2. In addition, calcium-binding proteins (i.e. S100 proteins), serine proteases, serine protease inhibitors (serpins), lipocalin and solute carriers were significantly affected by 13-cis RA25 In addition, Gene expression analysis in SEB-1 sebocytes and HaCaT keratinocytes with 72 hour 13-cis RA treatment. Revealed that there were changes in several genes involved in apoptosis and innate immunity such as TNFα-induced protein 2, TRAIL, interferon regulatory factor 1 (IRF1), interferon-induced proteins, NFκB, the death receptor, Fas and TIG3 (a.k.a. retinoic acid inducible gene 1 (RIG1)). TIG3 encodes an RNA helicase and represents a key intracellular protein that like the TLR3, can recognize viral double stranded RNA (dsRNA). 26 isotretinoin can inhebit cytokine storm thorough inhebtion of TLR-2 astudy demonstrated that treatment of patients with isotretinoin significantly decreased monocyte TLR-2 expression and subsequent inflammatory cytokine response to P. acnes after 1 week of therapy. This effect was sustained 6 months following cessation of therapy, indicating that TLR-2 modulation may be involved in the durable therapeutic response to isotretinoin.22 IN contrary, 13Cis retinoic Acid induced significant upregulation of toll-like receptor 3 (TLR3) , mitochondrial antiviral-signaling protein (MAVS) and retinoid-induced gene I (RIG-I) and IFN regulatory factor 1 expression in a time-dependent. 23 this can resulted in an immune response to dsRNA intermediate which can be partially generated during CoV-2 replicationTLR3 sensitized by dsRNA and cascades of signaling pathways (IRFs and NFκB activation, respectively) are activated to produce type I IFNs. The production of type I IFNs is important to enhance the release of antiviral proteins for the protection of uninfected cells. Sometimes, accessory proteins of CoV can interfere with TLR3 signaling and bind the dsRNA of CoV during replication to prevent TLR3 activation and evade the immune response. Interferon regulatory factor 1 (IRF1) was identified as a critical factor in mediating TRAIL induction by retinoic acid in NB4 APL leukemia cells and SK-BR-3 breast cancer cells. Interestingly, 13-cis RA significantly up-regulates IRF1 gene expression (2.42 fold increase) in SEB-1 sebocytes 27

Impact of antifungal drugs on inducing isotretinoin effect and concentration in targeted tissues

Itraconazole and fluconazole are triazole azole ring antifungal drugs, which are multiringed synthetic compounds containing three nitrogen atoms On the other hand, azole antifungal drugs have been demonstrated to inhibit cytochrome P450 28Thecytochrome P450 family (CYP26) enzymes are responsible for RA clearance, and are potential drug targets to increase concentrations of retinoid into targeted cells31 CYP26 Inhibitors Increases Retinoid Signaling in Intimal Smooth Muscle Cells32 Itraconazole has less inhibitive properties than the imidazoles in rat liver microsomes 29. ICZ interferes with the ergosterol synthesis pathway of the host cell and inhibits cytochrome P450 enzymes, particularly cyp 34 enzyme that metabolizes retinoic acid in human cells which increase retinoic acid concentration in to targeted mammalian cells40 leading to activation of TOLL-like receptors inducing its antiviral mechanism to induce type I IFN expression levels toward the induction of a preactivated state, thereby accelerating the virus-induced host cell response41 IFNs can serve as the first line of immune defense against viral infections.41 IFNs are very powerful cytokines, which play a key role in combatting pathogenic infections by controlling inflammation and immune response by directly inducing antipathogen molecular countermeasures.42There are three classes of IFNs: type I, type II, and type III.. Even though fluconazole has been shown to be a potent cytochrome P450 inhibitor 30 Here,we suggest that because antifungal drug. Fluconazol or itraconazol can inhibit cytochrome P450 enzymes, especially cype 26 which control retinoic acid concentration into human cells antifungal can enhance both isotretinoin effect and Concentrations in Target Tissues This in turn lead to hyper interferon induction and synthesis in case of COVID-19 Astudy found that fluconazole has been shown to be a potent cytochrome P450 inhibitor32 Safety of Aerosolized Isotretinoin Isotretinoin (Accutane, Roche Laboratories Inc, Nutley, NJ) is an important drug, not only for the treatment of severe acne, but also for other diagnoses and in chemoprevention settings. Because the use of isotretinoin is increasing, it is important for physicians to be aware of the adverse events, toxicities, and management issues related to its use. The most important issue is that of congenital defects, which has resulted in new pregnancy prevention policies and programs implemented by the manufacturer. A relatively new concern is that of depression associated with isotretinoin use, also resulting in new policies placed by the manufacturer and the FDA., But here, in our review we highly recommend that any researcher who wants to apply isotritinoin clinically covid-19 his clinical study must be a small pilot study investigating whether there is any efficacy signal that warrants a larger Phase 2B trial, or any harm that suggests that such a trial should not be done. The investigator will examine all of the biologic, physiological, and clinical data to determine whether a Phase 2B trial is warranted. And he also must abide by these rules :Isotretinoin must be give in the form of aerosol thorough respiratory route in order for it to has an effect that is focused only on lung cells so as not to affect any other organs. Aerosol inhalation can deposit drug directly on the population of cells caught up in the early phase of cancer, potentially achieving much more efficiency compared with reliance on diffusion from the blood. Direct application of aerosolized retinoic acid to the lung epithelium may avoid much of the protein binding, and serious side effects on the other organs especially, congenital organs thus greatly increasing potency at the target site.35 Because a study on rabbits demonstrated that isotretinoin can be given in the form of aerosol without serious side effects . Repeated high doses of 13 cis retinoic by inhalation resulted in moderate loss of body weight, but microscopic investigation of ten tissues inhalation rout without any damage in lung including lung and oesophagus did not detect any significant aerosol-induced damage therefore inhaled isotretinoin might provide sufficient drug to the target cells in lung for efficacy while avoiding systemic toxicity © 2000 Cancer Research Campaign33 In 2006, a clinical trial conducted to assess the feasibility of retinoids for the treatment of emphysema, the FORTE study, was published (NCT00000621)33. In that study, 148 patients from five university hospitals were recruited and randomized to receive ATRA at either low dose (1 mg/kg/day for 4 days/wk) or high dose (2 mg/kg/day for 4 days/wk), 13-cis retinoic acid (1 mg/kg/day, daily), or placebo for 6 months, followed by a 3-month crossover phase. Subsequently, they were observed for an additional 9 months before the final assessment. In the trial, retinoids(13 cis retinoic acid ) were proven to be safe as the drug-related AEs were generally mild.37 In addition, aerosolized isotretinoin must be given with low dose in accordance to patient weight and also it must be given gradually concentration thorough a short period not exceeding 14 days from the date of giving the first dose In contrast to the long course of treatment, which is considered chronic treatment and Aerosolized 13 cis retinoic acid must be be given gradually in one daily dose increases from 0.2 mg/kg/day to 2 mg/kg/day as inhaled 13 cis retinoic acid therapy for 14 days A study demonstrated that the application of aerosolized retinoic acid system led to a rise of Retinoic Acid levels in lung, but not liver or plasma. Cellular lung levels of retinol, retinyl palmitate, and retinyl stearate also appeared to be unaffected (245.6 ± 10.7, 47.4 ± 3.4, and 132.8 ± 7.7 ng•g-1 wet weight, respectively). And also demonstrated that the application of this aerosolized Retinoic Acid also induced a dose-dependent protein expression of the cellular retinol-binding protein 1 (CRBP-1) in lung, without apparent harmful side effects.38 Although, more than one clinical study reported safety and non serious side effects of systemic isotretinon but we highly recommend that isotretinoin must be given in the form of aerosol with short period of tratment and with low gradual dose to target lung cells only for avoiding any potential side effects. A clinical study applied on 1166 patients thorough phase III trial (NCI #I91-0001) at a National Cancer Institute (NCI) demonstrated that after the median follow-up of 3.5 years, there were no statistically significant differences between the placebo and isotretinoin arms with respect to the time to SPTs, recurrences, or mortality. In this study Patients were randomly assigned to receive a placebo or the retinoid isotretinoin (30 mg/day) for 3 years in a double-blind fashion. Patients were stratified at randomization by tumor stage, histology, and smoking status. The primary endpoint (time to SPT) and the secondary endpoints (times to recurrence and death) were analyzed by log-rank test and the Cox proportional hazards model. All statistical tests were two-sided.34 A study conducted on 720 patients who had received one or more courses of oral isotretinoin treatment, and had a mean follow up period of 4.9 years (range 2/12 years). Most patients (442) had received a total cumulative dose of 120/200 mg/kg body weight. One hundred and sixty two patients received a cumulative dose of <120 mg/kg body weight, and 116 received a cumulative dose <200 mg/kg. Finally this study proved that oral isotretinoin in the treatment of acne is a safe drug, with no serious long term side effects.36

Safety of Aerosolized fluconazole

A study demonstrated that fluconazole can be given via route of inhalation. Respiratory fungal diseases therapy is still facing challenges as a result of increasing autoimmune disorders, cancers, and immunosuppressive medication usage. Fluconazole is a wide spectrum antifungal agent and is still used successfully in the treatment of opportunistic infections in combination with other antifungal agents. Since, the treatment of respiratory fungal diseases requires prolonged hospitalization; it may increase the chances of other opportunistic infections. Considering the reported drug resistance and adverse effects of systemic administration, it appears that localized pulmonary antifungal therapy may be a suitable alternative route. According to the reported suitable inhalation properties of spray dried powders; spray drying technique was used to prepare fluconazole powders.39

ELIGIBILITY:
Inclusion Criteria:

* Adult SARI patients with 2019-ncov infection confirmed by PCR;
* Absolute value of lymphocytes < 0. 6x 109/L;
* Severe respiratory failure within 48 hours and requires admission to ICU. (severe respiratory failure was defined as PaO2/FiO2 < 200 mmHg and was supported by positive pressure mechanical ventilation (including non-invasive and invasive mechanical ventilation, PEEP>=5cmH2O))

Exclusion Criteria:

* Age < 18
* Pregnant
* Allergic to experimental drugs
* The underlying disease is very serious and the expected survival time is less than 6 months (such as advanced malignant tumor);
* COPD or end-stage lung disease requires home oxygen therapy
* Expected survival time not exceeding 48 hours
* Participated in other clinical intervention trials within the last 3 months
* Autoimmune diseases
* A history of organ, bone marrow or hematopoietic stem cell transplantation
* Received radiotherapy and chemotherapy for malignant tumor within 6 months
* HIV infected patients or diagnosed with acquired immunodeficiency within the past year (CD4 T cells <=200/mm3)
* Patients receiving anti-hcv treatment
* 90 days of retinal detachment or eye surgery
* Permanent blindness in one eye
* History of iritis, endophthalmitis, scleral inflammation or retinitis
* The competent physician considered it inappropriate to participate in the study

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2020-10-20 (Estimated); Primary Completion 2020-11-20 (Estimated); Study Completion 2020-11-20 (Estimated)

PRIMARY OUTCOMES:
lung injury score | at 7and 14 days
  proportion of lung injury score decreased or increased after treatment

SECONDARY OUTCOMES:
Absolute lymphocyte counts | at day 7 and 14 after randimization
  Lymphocyte counts
Serum levels of CRP, ESR ,IL-1,IL-6,TNF and Type I interferons | at day 7 and 14 after randimization
  Serum levels of CRP, ESR ,IL-1,IL-6,TNF and Type I interferons
All cause mortality rate | at day 7 and 14
  Died
Serum level of viral RNA | at day 7 and 14
  Serum level of viral RNA
Ventilation free days | at 14 days
  Ventilation free days
ICU free days | at 14 days
  ICU free days

CONTACTS AND LOCATIONS:
Overall Officials: mahmoud Elkazzaz, B.Sc of biochemistry, Principal Investigator — Faculty of Science,Damietta university
Locations (1):
- Kafr El-sheikh University, Cairo, Kafr el-Sheikh Governorate, Egypt